CLINICAL TRIAL: NCT06654518
Title: The Prognostic Accuracy of Bone Density and Alveolar Ridge Width Estimated by CBCT in Predicting Primary Implant Stability: Clinical Study.
Brief Title: Prediction of Primary Dental Implant Stability Preoperatively Using CBCT of the Planned Implant Site.
Acronym: CBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, lecturer of oral and maxillofacial surgery department, Faculty of dentistry, Mansoura university, Egypt., Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A28030123
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2024-10

CONDITIONS: Prediction of Primary Implant Stability From Bone Quality Obtained Prior to Implant Placement Using CBCT
Keywords: bone density, alveolar ridge width, insertion torque, resonance frequency analysis
MeSH Terms: interventions — Bone Density

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants underwent preoperative CBCT measurements to guide the dental implant placement process. (Experimental): Participants in this arm underwent preoperative Cone Beam Computed Tomography (CBCT) scans to assess bone density and alveolar ridge width. The data obtained from these scans was used to guide dental implant placement, with the primary goal of predicting the primary stability of the implant. The intervention involved using CBCT technology to gather precise anatomical details that help optimize implant placement and ensure adequate bone support for the implant.
  Interventions: Diagnostic Test: Preoperative CBCT for Bone Density and Ridge Width Measurement

INTERVENTIONS:
Diagnostic Test: Preoperative CBCT for Bone Density and Ridge Width Measurement — Participants in this arm underwent preoperative Cone Beam Computed Tomography (CBCT) scanning to evaluate bone density and alveolar ridge width. The CBCT scans provide high-resolution, 3D images, which was used to guide the planning and placement of dental implants. The primary goal of the intervention was to assess how well the measurements obtained from CBCT could predict the primary stability of the implants postoperatively.

SUMMARY:
This study aimed to assess whether preoperative characteristics of the implant site, such as bone density and alveolar ridge width, assessed using cone beam computed tomography (CBCT), are significantly associated with primary stability, as assessed by resonance frequency analysis (RFA) and final insertion torque value (ITV), and thereby investigate if it is feasible to predict primary stability preoperatively using this form of radiologic examination of the planned implant site. All patients underwent preoperative CBCT. The bone density and alveolar ridge width were assessed. The primary implant stability quotient (ISQ) values were assessed by a wireless magnetic-based Osstell ISQ RF Analyzer.

DETAILED DESCRIPTION:
The quality and quantity of bone available for placing dental implants are key factors in the success of these implants. Implants placed in bone with insufficient quantity or poor quality have a higher risk of failure. As a result, evaluating the bone structure prior to implant placement surgery is essential for proper planning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be free from any systemic conditions that would contraindicate dental implant surgery.
2. Good oral hygiene.
3. Age above 18 years.
4. The planned implant site must have sufficient alveolar bone volume.

Exclusion Criteria:

1. Patients who have undergone radiation therapy to the head and neck region within the last 12 months.
2. Uncontrolled diabetes.
3. Patients who underwent dental extractions or bone augmentation at the planned implant site during the last six months in order to guarantee uniform bone maturation.
4. Severe clenching or bruxism is present.
5. Acute infection at the planned implant site.
6. Implant sites requiring a procedure for bone gain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Primary Implant Stability Using Resonance Frequency Analysis (RFA)and final insertion torque value (ITV) | Measured immediately after implant placement
  The primary outcome measure was the primary stability of the dental implants as determined by resonance frequency analysis (RFA) and final insertion torque value (ITV). The Implant Stability Quotient (ISQ) was measured immediately after the implant placement. ITV and ISQ values were corelated with the preoperative CBCT measurements of bone density and alveolar ridge width to evaluate the prognostic accuracy of CBCT in predicting primary implant stability.

CONTACTS AND LOCATIONS:
Overall Officials: Soaad T Badawi, Lecturer, Oral Surgery, MU, Principal Investigator — Faculty of dentistry, Mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
"Individual Participant Data (IPD) from this study will not be shared due to privacy and confidentiality concerns, as well as institutional policies that restrict the sharing of sensitive personal data. The data collected includes health-related information that must be protected according to ethical guidelines and local regulations."

REFERENCES:
- [Background] de Elio Oliveros J, Del Canto Diaz A, Del Canto Diaz M, Orea CJ, Del Canto Pingarron M, Calvo JS. Alveolar Bone Density and Width Affect Primary Implant Stability. J Oral Implantol. 2020 Aug 1;46(4):389-395. doi: 10.1563/aaid-joi-D-19-00028. PMID 32221558